CLINICAL TRIAL: NCT06563518
Title: The Clinical Investigation of Toothpaste Containing Zinc Lactate as Compared to Colgate Cavity Protection Toothpaste in Reducing Plaque and Gingivitis - a Six-month Study in Thailand
Brief Title: Clinical Study of Toothpaste Containing Zinc Lactate as Compared to Colgate Cavity Protection Toothpaste.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRO-2021-10-PGN-MRO-YPZ
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Gingivitis; Plaque
MeSH Terms: conditions — Gingivitis; Plaque, Amyloid | interventions — Meridol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group 1 (Experimental): Toothpaste
  Interventions: Drug: Meridol
- Group II (Active Comparator): Toothpaste
  Interventions: Drug: Colgate Cavity Protection

INTERVENTIONS:
Drug: Meridol — toothpaste
  Arms: Group 1
Drug: Colgate Cavity Protection — toothpaste
  Arms: Group II

SUMMARY:
The objective of this six-month clinical research study is to evaluate the clinical efficacy of two dentifrices - Toothpaste containing zinc lactate and Colgate Cavity Protection Toothpaste in reducing gingivitis and dental plaque in adults.

ELIGIBILITY:
Inclusion Criteria:

* Subjects, ages 18-70, inclusive.
* Availability for the six-month duration of the clinical research study.
* Good general health.
* Minimum of 20 uncrowned permanent natural teeth (excluding third molars).
* Initial gingivitis index of at least 1.0 as determined by the use of the Loe and Silness Gingival Index.
* Initial plaque index of at least 1.5 as determined by the use of the Quigley and Hein Plaque Index (Turesky Modification).
* Signed Informed Consent Form

Exclusion Criteria:

* Presence of orthodontic bands.
* Presence of partial removable dentures.
* Tumor(s) of the soft or hard tissues of the oral cavity.
* Advanced periodontal disease (purulent exudate, tooth mobility, and/or extensive loss of periodontal attachment or alveolar bone).
* Five or more carious lesions requiring immediate restorative treatment.
* Antibiotic use any time during the one-month period prior to entry into the study.
* Participation in any other clinical study or test panel within the one month prior to entry into the study.
* Dental prophylaxis during the past two weeks prior to baseline examinations.
* History of allergies to oral care/personal care consumer products or their ingredients.
* On any prescription medicines that might interfere with the study outcome.
* An existing medical condition that prohibits eating or drinking for periods up to 4 hours.
* History of alcohol or drug abuse.
* Pregnant or lactating subjects.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2022-07-10 (Actual); Study Completion 2022-07-10 (Actual)

PRIMARY OUTCOMES:
Gingivitis Assessment | baseline, 3 months and 6 months
  A Loe-Silness Gingival Index score from 0 to 3 will be assigned by the examining dentist to all scoreable surfaces of the maxillary and mandibular teeth using a dental light and dental mirror.
Plaque Assessment | baseline, 3 months and 6 months
  A Quigley-Hein Plaque Index score of 0 to 5 will be assigned to all scoreable disclosed surfaces of the maxillary and mandibular teeth using a dental light and dental mirror

CONTACTS AND LOCATIONS:
Overall Officials: Terdphong Triratana, Principal Investigator — Managing Director of Dental Research Center
Locations (1):
- Mahidol University, Ratchathewi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Seriwatanachai D, Triratana T, Kraivaphan P, Huber N, Poth T, Mateo LR, Stellitano M, Zhang YP. Effectiveness of a novel amine + zinc + fluoride toothpaste in reducing plaque and gingivitis: results of a six-month randomized controlled trial. BMC Oral Health. 2025 Feb 5;25(1):188. doi: 10.1186/s12903-025-05551-z. PMID 39910536